CLINICAL TRIAL: NCT06790264
Title: Exploring the Tumor Micro-Environment with 68Ga-FAPi-46 PET/CT in Breast Cancer. a Phase II Study to Evaluate the Comparison of 68Ga-FAPi-46 and 18F-FDG Uptake in Patients with Different Breast Cancer Subtypes
Brief Title: Exploring the Tumor Micro-Environment with 68Ga-FAPi-46 PET/CT in Breast Cancer
Acronym: FAPI-PET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UID 4047
Record Dates: First submitted 2025-01-17; First posted 2025-01-24 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Invasive; Node Positive Breast Cancer
Keywords: 68Ga-FAPi-46 PET/CT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-FAPi-46 PET/CT (Experimental): Study participants will undergo baseline assessments at enrollment with 68Ga-FAPi-46 PET/CT
  Interventions: Procedure: 68Ga-FAPi-46 PET/CT

INTERVENTIONS:
Procedure: 68Ga-FAPi-46 PET/CT — Study participants will undergo baseline assessments at enrollment with 68Ga-FAPi-46 PET/CT

SUMMARY:
This study is a prospective, non-interventional, open-label study to evaluate the glucose metabolism and the expression of the imaging agent 68 Gallium-Fibroblast Activation Protein Inhibitor-46 (68Ga-FAPi-46) with PET imaging, in woman affected by Breast Cancer (BC) and referred to diagnostic imaging work-up prior to primary therapy.

DETAILED DESCRIPTION:
All patients affected by newly diagnosed, clinically N-positive BC that have already undergone a baseline 2-deoxy-2-[fluorine-18]fluoro-D-glucose (18F-FDG) PET/CT (T1) will be screened for eligibility. Patients who will meet all inclusion/exclusion criteria will be considered eligible and asked to participate to the study after signing the informed consent form. Patients' eligibility will be evaluated by the referent nuclear medicine physician (T2). Considering the clinical experience of the investigators, we expect to complete patient enrolment in 12 months after study accrual

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, biopsy proven breast cancer;
* Diagnosis of invasive breast cancer;
* Tumor diameter more than 2 centimeters;
* Radiological evidence of axillary nodes involvement;
* 18F-FDG PET/CT performed as baseline diagnostic procedure, during routine diagnostic work-up;
* 68Ga-FAPi-46 PET/CT performed within 4 weeks from 18F-FDG PET/CT;
* Patients suitable to primary treatment (surgery or neo-adjuvant therapy);
* 68Ga-FAPi-46 PET/CT performed within 8 weeks from primary treatment;
* Female patients;
* Age ≥18;
* Willing to sign informed consent form.

Exclusion Criteria:

* Pregnant or nursing patients;
* Unable to stay flat and cannot tolerate PET scan;
* Sample tissue from biopsy unavailable for assessing Fibroblast Activation Protein (FAP) expression;
* Eastern Cooperative Oncology Group (ECOG) performance status ≥2.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Comparison of 68Ga-FAPi PET/CT and 18F-FDG PET/CT positivity rate | 3 months
  Comparison of 68Ga-FAPi PET/CT and 18F-FDG PET/CT of positivity rate (percentage of detection of metastatic patients)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Ceci, MD, Principal Investigator — European Istitute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No